CLINICAL TRIAL: NCT03793088
Title: xCures/CancerCommons Enhanced Learning Treatment Selection and Analysis With Outcomes Research (XCELSIOR) Study: A Patient-Centric Platform Trial for Precision Oncology
Brief Title: A Patient-Centric Platform Trial for Precision Oncology
Acronym: XCELSIOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: xCures (Industry)
Collaborators: Cancer Commons (Other); Musella Foundation for Brain Tumor Research and Information, Inc. (Unknown); Pediatric Oncology Experimental Therapeutics Investigators Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: XC3-GCTA-2018
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Oncology
Keywords: Glioblastoma; Glioma; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Neoplasms; Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
XCELSIOR is a non-interventional data registry. Information about treatments, treatment decisions and rationale, and patient outcomes including safety and effectiveness of anti-cancer therapy and associated supportive care will be collected for analysis.

DETAILED DESCRIPTION:
XCELSIOR is patient-centric study for the registration of cancer patients, operations of a virtual tumor board, insight capture in clinical decision making, and collection of longitudinal, observational data in a cancer registry. Patient intake into XCELSIOR will occur through the Cancer Commons Web portal. This includes consent to participate in the data registry, including the collection and review of medical information by a Virtual Tumor Board, generation of patient-specific treatment options with supporting rationale, access to treatment access support services, and inclusion into a registry study that includes safety and efficacy outcomes tracking. Patients will be treated and tracked in their original treatment setting and the data generated will form part of a systematic framework combining expert judgment with artificial intelligence to maximize information gain and improve treatment option set development for individual cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients with known or suspected recalcitrant or advanced cancer are eligible to enroll through the Cancer Commons Website
* Patients with any performance status, comorbidity or disease severity are eligible
* Patients or their legally-authorized representative must be willing and able to provide written, informed consent (and assent, if applicable)

Exclusion Criteria:

* Patients must be a resident of or receiving care within the United States or US territories.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will initially include up to 10,000 adult and pediatric patients with recalcitrant or advanced cancers.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 5 Years
Overall Survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Shapiro, Principal Investigator — xCures / Cancer Commons
Locations (1):
- Cancer Commons, Los Altos, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Cancer Commons Website — https://www.cancercommons.org/
- See also: xCures Website — https://www.xcures.com/patients/

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03793088/Prot_ICF_000.pdf